CLINICAL TRIAL: NCT06984952
Title: Effectiveness of Enhanced Recovery After Surgery (ERAS) on Postoperative Recovery After Minimally Invasive Gastrectomy: A Multi-center Open-labeled Randomized Controlled Study
Brief Title: Effectiveness of ERAS on Postoperative Recovery After Minimally Invasive Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); Severance Hospital (Other); Chungnam National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); National Cancer Center, Korea (Other Government); The Catholic University of Korea (Other); Ajou University School of Medicine (Other); Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2501-115-1609
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Enhanced Recovery After Surgery; Gastrectomy for Gastric Cancer
Keywords: enhanced recovery after surgery; stomach neoplasms; gastrectomy for gastric cancer; pain, postoperative
MeSH Terms: conditions — Stomach Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A prospective randomized open-labeled, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Perioperative care for minimally-invasive gastrectomy is managed according to ERAS protocol.
  Interventions: Procedure: ERAS protocol
- Conventional group (No Intervention): Perioperative care for minimally-invasive gastrectomy is managed according to our current perioperative practice

INTERVENTIONS:
Procedure: ERAS protocol — The ERAS protocol includes pre-admission patient education through audiovisual materials; reduction of perioperative fasting duration with preoperative carbohydrate loading and early postoperative oral intake; multimodal prophylaxis for postoperative nausea and vomiting; early removal of surgical drains and intravenous lines; early mobilization; and multimodal analgesia aimed at minimizing postoperative opioid use. The detailed protocol used in this study has been published previously [https://doi.org/10.5230/jgc.2025.25.e27].
  Arms: ERAS group

SUMMARY:
This prospective, randomized, open-label, multicenter study is designed to evaluate the impact of an enhanced recovery after surgery (ERAS) protocol on the rate of meeting discharge criteria in patients undergoing minimally-invasive gastrectomy for gastric cancer. We hypothesize that implementation of our ERAS protocol will significantly increase the proportion of patients who meet standardized discharge criteria following minimally-invasive gastrectomy.

DETAILED DESCRIPTION:
Adult patients undergoing elective minimally invasive gastrectomy were randomly allocated to receive either the ERAS protocol (n = 154) or the conventional protocol (n = 154). The conventional group received the current standard perioperative care at our institution, whereas the ERAS group received a newly developed ERAS protocol, which included preoperative carbohydrate loading, reduced perioperative fasting duration, and multimodal opioid-sparing analgesia. The primary outcome was the proportion of patients who met standardized discharge criteria at 9:00 AM on postoperative day 4. Secondary outcomes included the EQ-5D-5L index assessed at 24, 48, 72, and 96 hours postoperatively; pain intensity at rest and during coughing measured using an 11-point numeric rating scale at 2, 24, 48, and 72 hours postoperatively; gastrointestinal dysfunction assessed using the I-FEED score at 24, 48, and 72 hours postoperatively; the incidence of postoperative nausea and vomiting within 0-24, 24-48, and 48-72 hours after surgery; the incidence of major postoperative complications classified by the Clavien-Dindo grading system during hospitalization; and postoperative length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years scheduled to undergo elective laparoscopic or robotic gastrectomy for gastric cancer
* American Society of Anesthesiologists physical status classification I to III
* Ability to provide written informed consent, demonstrate understanding of the study protocol, and complete patient-reported outcome measures appropriately

Exclusion Criteria:

* Requirement for resection of organs other than the stomach during surgery (except for cholecystectomy)
* History of upper abdominal surgery (except for cholecystectomy)
* Known hypersensitivity to fentanyl, ropivacaine, acetaminophen, or non-steroidal anti-inflammatory drugs
* Determined by the investigator or study personnel to be otherwise unsuitable for participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who fulfilled all of the predefined discharge criteria | At 9:00 AM on postoperative day
  Discharge criteria were defined as meeting all of the following conditions:
  * Tolerance of a soft blended diet (SBD) for at least 24 hours
  * Unaided ambulation of at least 600 meters
  * Adequate pain control, defined as a numeric rating scale (NRS) score of ≤ 3, achieved with oral non-opioid analgesics
  * Absence of abnormal physical examination findings or laboratory test results

SECONDARY OUTCOMES:
Postoperative pain score | postoperative 2, 24, 48, and 72 hours
  11-pointed NRS pain score at resting/coughing NRS (0-10): 0,"no pain"; 10, "worst pain imaginable"
Postoperative gastrointestinal dysfunction | postoperative 24, 48, and 72 hours
  I-FEED score 3 points or more (postoperative gastrointestinal intolerance and dysfunction)
Postoperative nausea and vomiting | From the end of surgery to 24, 48, and 72 hours postoperatively
  Incidence of postoperative nausea and vomiting (%)
Quality of recovery assessed using the EQ-5D-5L questionnaire | postoperative 24, 48, and 72 hours
  EQ-5D-5L index scores are calculated from the EQ-5D-5L questionnaire using the Korean value set validated for the Korean population. (range: 0 to 1.000, with higher scores indicating better recovery) (Kim SH, Ahn J, Ock M, et al. The EQ-5D-5L valuation study in Korea. Qual Life Res. 2016; 25: 1845-1852)
Major postoperative complication | At 30 days postoperatively
  Major postoperative complications are defined as events classified as Clavien-Dindo grade IIIa or higher and are assessed based on their incidence within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Do Joong Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (10):
- South Korea (10):
  - Pusan National University Hospital, Busan
  - Dongsan Hospital, Keimyung University School of Medicine, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance hospital, Seoul
  - SMG-SNU Boramae Medical Center,, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee HJ, Kim J, Koo BW, Suh YS, Lee JM, Han DS, Hong SH, Lee HH, Yoo YC, Kim HI, Rho JY, Yoon HM, Kim HY, Hur H, Kim HJ, Choi CI, Hong B, Lee SI, Park K, Ryu SW, Park DJ. Survey of Perioperative Practices in Gastric Cancer Surgery for Establishing an Enhanced Recovery After Surgery Program Across 10 Tertiary Hospitals in South Korea. J Gastric Cancer. 2025 Jul;25(3):424-436. doi: 10.5230/jgc.2025.25.e27. PMID 40631472
- [Background] Lee HJ, Kim J, Yoon SH, Kong SH, Kim WH, Park DJ, Lee HJ, Yang HK. Effectiveness of ERAS program on postoperative recovery after gastric cancer surgery: a randomized clinical trial. Int J Surg. 2025 May 1;111(5):3306-3313. doi: 10.1097/JS9.0000000000002328. PMID 40072360